CLINICAL TRIAL: NCT01070693
Title: Randomized Clinical Trial of Lichtenstein Patch or Prolene Hernia System for Inguinal Hernia Repair
Brief Title: Lichtenstein Patch or Prolene Hernia System (PHS) for Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jaana Vironen, Consultant, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TYH1333
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Pain
Keywords: Inguinal hernia; Open mesh repair; Long term outcome; Recurrence; Discomfort
MeSH Terms: conditions — Chronic Pain; Hernia, Inguinal; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolene Hernia System device (Experimental): Inguinal hernia repair either with a bilayer mesh (PHS)
  Interventions: Procedure: Open mesh inguinal hernia repair; Device: Prolene Hernia System
- Lichtenstein (Experimental): Inguinal hernia repair with the Lichtenstein technique
  Interventions: Procedure: Open mesh inguinal hernia repair; Procedure: Lichtenstein technique

INTERVENTIONS:
Procedure: Open mesh inguinal hernia repair — Inguinal hernia repair either with the bilayer mesh or the Lichtenstein technique
Device: Prolene Hernia System — Prolene Hernia System
  Arms: Prolene Hernia System device
Procedure: Lichtenstein technique — Lichtenstein technique
  Arms: Lichtenstein

SUMMARY:
This randomised prospective study was designed to compare the convalescence and the long-term sequelae in inguinal hernia repair with either a bilayer mesh as devised by Gilbert (Prolene Hernia System®) or an onlay mesh applied according to Lichtenstein.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral
* Primary or recurrent

Exclusion Criteria:

* body-mass index over 40kg/m2, severe co-morbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2001-09; Primary Completion 2005-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Central Hospital, Espoo, Finland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Included were 300 adult patients (282 men, 18 women) referred for elective repair having unilateral or bilateral inguinal hernias. Study period: September 2001 - January 2004, outpatient unit of Jorvi Hospital (Helsinki University Central Hospital, Espoo, Finland).
Period: Overall Study
Arm/Group | Prolene Hernia System Device | Lichtenstein
Started | 150 | 149
Completed | 122 | 110
Not Completed | 28 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolene Hernia System Device | Lichtenstein | Total
Number analyzed (Participants) | 150 | 149 | 299
Age, Continuous [Median (Full Range); unit: years] | 46 [19 to 72] | 47 [20 to 70] | 46 [19 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 140 | 141 | 281
Region of Enrollment [Number; unit: participants]
  Finland | 150 | 149 | 299

OUTCOME MEASURES:

1. Primary Outcome: Long-term Sequelae
Description: Any pain at five years
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Prolene Hernia System Device | Lichtenstein
Number analyzed (Participants) | 122 | 110
percentage of participants | 10 | 13

ADVERSE EVENTS:
Arm/Group | Prolene Hernia System Device | Lichtenstein
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/149
Other Adverse Events (participants affected / at risk) | 0/150 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No